CLINICAL TRIAL: NCT05811182
Title: Prospective Analysis of the Correlation Between Hyperreflective Dots in the Vitreous Body and the Appearance of a Pseudophakic Cystoid Macular Edema
Brief Title: Vitreous Hyper Reflective Dots in Association With Pseudophakic Cystoid Macular Edema
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 30-273 ex 17/18
Record Dates: First submitted 2023-03-01; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cystoid Macular Edema Following Cataract Surgery; Vitreous Hyperreflective Dots
Keywords: VHD; phacoemulsification; CME

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the association between vitreous hyper-reflective dots (VHD) and the macular thickness changes following uneventful phacoemulsification. In this prospective study the investigators performed optical coherence tomography (OCT) imaging in patients undergoing cataract surgery preoperatively and postoperatively after 1 week, 1 month and 3 months and analyzed the OCTs for VHDs. The investigators then measured the macular thickness in patients with VHDs and without VHDs and correlated the macular thickness with the number of VHDs.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cataract surgery
* minimum age 18 years
* phacoemulsification technique
* subsequent implantation of a monofocal hydrophobic acrylic intraocular lens

Exclusion Criteria:

* intraoperative complications including capsule rupture with or without anterior vitrectomy
* iris bites
* previous interventions including vitrectomy
* glaucoma surgery
* exudative or dry age-related macular degeneration
* presence of diabetes
* history or presence of retinal vein occlusion or uveitis
* epiretinal glioses

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cataract surgery using the manual anterior continuous curvilinear capsulorhexis phacoemulsification technique for the removal of the crystalline lens and subsequent implantation of a monofocal hydrophobic acrylic intraocular lens in the capsular bag
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
vitreous hyperreflective dots | preoperatively until 3 months postoperatively
  Change of correlation between occurrence of vitreous hyperreflective dots and the macular thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria